CLINICAL TRIAL: NCT04879953
Title: Effect of Pressurised Intraperitoneal Aerosol Chemotherapy on the Survival Rate of Patients With Peritoneal Carcinomatosis of Gastric Origin
Brief Title: Effect of the PIPAC on the Survival Rate of Patients With Peritoneal Carcinomatosis of Gastric Origin
Status: Completed | Type: Observational
Sponsor: Association Francaise de Chirurgie (Other)
Responsible Party: Principal Investigator, Pr Catherine Arvieux, Professeur, Association Francaise de Chirurgie
Other Study IDs: PIPAC
Record Dates: First submitted 2021-05-05; First posted 2021-05-10 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Carcinomatosis, Peritoneal
MeSH Terms: conditions — Peritoneal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PIPAC CHEM: PIPAC associated with systemic chemotherapy
  Interventions: Drug: PIPAC with systemic chemotherapy
- ONLY CHEM: systemic chemotherapy alone
  Interventions: Drug: Systemic chemotherapy alone

INTERVENTIONS:
Drug: PIPAC with systemic chemotherapy — PIPAC procedures were performed every 6 to 8 weeks, alternating with systemic chemotherapy, replacing a cycle of intravenous chemotherapy.
  Groups: PIPAC CHEM
Drug: Systemic chemotherapy alone — Intravenous chemotherapy
  Groups: ONLY CHEM

SUMMARY:
Pressurised intraperitoneal aerosol chemotherapy is a new surgical technique, developed for the treatment of initially unresectable peritoneal carcinomatosis. The objective of this study was to compare the results of PIPAC associated with systemic chemotherapy with those of systemic chemotherapy alone in patients with gastric peritoneal carcinomatosis without metastasis other than peritoneal, and WHO performance status <3.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or over
* Patients with adenocarcinoma-type gastric non-resectable péritonéale carcinomatosis.
* Patients without metastasis other than peritoneal.
* WHO performance status <3
* Patients treated either with PIPAC administered in alternation with systemic chemotherapy (PIPAC_CHEM) or by systemic chemotherapy alone (ONLY_CHEM)
* Patient informed

Exclusion Criteria:

- Patients opposed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of adult patients with adenocarcinoma-type gastric non-resectable PC, without metastasis other than peritoneal, treated either with PIPAC administered in alternation with systemic chemotherapy or by systemic chemotherapy alone. All patients receiving PIPAC in our hospital during the study period were included. The patients in the group had been treated during the same period and were carefully selected according to age, general state of health (WHO performance status <3) and absence of extra-peritoneal metastases so as to match as closely as possible the patients in the PIPAC group.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Overall survival at 6 months | 6 months
  Overall survival at 6 months from diagnosis of carcinomatosis

SECONDARY OUTCOMES:
Duration of hospital stay | 6 months
  duration of hospitalization up to 6 months after the diagnosis of carcinomatosis
overall survival from the diagnosis of carcinomatosis and from the diagnosis of the primary tumour. | 3 years
  overall survival throughout the study follow-up from the diagnosis of carcinomatosis and from the diagnosis of the primary tumour.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Arvieux, Principal Investigator — Grenoble Hospital
Locations (1):
- CHUGA, Grenoble, France